CLINICAL TRIAL: NCT03098329
Title: A New Approach to Controlling Chlamydia Transmission in Young People
Brief Title: Check it: A New Approach to Controlling Chlamydia Transmission in Young People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Patricia Kissinger, Principal Investigator, Tulane University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 16-964337; 1R01HD086794-01A1 (NIH)
Record Dates: First submitted 2017-03-14; First posted 2017-03-31 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Chlamydia Trachomatis Infection; Gonorrhea
Keywords: Screening; men; expedited treatment
MeSH Terms: conditions — Gonorrhea; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: Community based screening of young men for chlamydia and gonorrhea, expedited treatment for positive subjects and their sexual partners
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ct/GC screening (Experimental): Community screening of men for Ct and GC is not normally done. We are testing to see if this intervention will impact the rates of Ct and GC among women
  Interventions: Other: Ct/GC screening

INTERVENTIONS:
Other: Ct/GC screening — Men aged 15-26 years old will be tested for chlamydia and gonorrhea at community based venues; positive men and their sexual partners will be offered expedited treatment at participating pharmacies; positive men will be asked to be rescreened for Ct/GC at 3 months post treatment.

SUMMARY:
This study, named "Check it," is a bundled program for African American (AA) men ages 15-24 that includes community testing for chlamydia and gonorrhea, expedited treatment for subjects who test positive and their female sexual contacts, and rescreening for these two sexually transmitted infections.

DETAILED DESCRIPTION:
Participants (N=4854) will be recruited through community partners, at events and using social marketing campaigns including advertisements, referrals from other participants, social media, and a web based educational website (Web-Ed). After establishing eligibility, written informed consent will be obtained. Subjects will complete a survey and provide a urine specimen for chlamydia (Ct) and gonorrhea (GC) testing and will provide their preferred contact information in order to be contacted about their test results. The testing laboratory will report positive results per LA hygiene code LAC 51:II.105: http://ldh.la.gov/assets/oph/Center-PHCH/Center-CH/infectious-epi/Surveillance/sanitarycode.pdf. Tulane study staff will contact participants to inform them of their results. If the participant tests positive for Ct and/or GC, the subject will be offered expedited treatment for the subject and the subject's recent sex partners. The subject may choose to pick up medication at a local pharmacy or medication can be mailed to the subject. Staff will also ask the participant to contact his partner(s) and provide them with the Check It staff's contact information so that staff can let the partner know that they have been exposed to an infection and offer the subject's sexual partner expedited treatment options if the participant did not already provide the subject's sexual partners with that information. No information provided by the participant will be shared with his partners. The study will cover the cost of the medications for subjects who test positive for either or both organisms and their sexual partners. Three months after treatment, male subjects who were positive will be asked to be re-screened and if positive, staff will conduct similar expedited treatment and partner services. Any subject who provides consent for annual testing reminders will be reminded using their preferred method of contact.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as African American or Black
* Identifies as male
* 15-26 years of age
* Lives or spends most of his time in Orleans Parish
* Had vaginal sex with at least one woman
* Has not taken azithromycin in the past 7 days

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Unable to speak or understand English
* Previously enrolled in the study by self-report

Ages: 15 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Identifies as male
Enrollment: 1907 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Rate of chlamydia in women | up to 60 months
  primary outcome

SECONDARY OUTCOMES:
Rate of gonorrhea in women | up to 60 months
  secondary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Tulane University School of Public Health and Tropical Medicine, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Campbell MB, Ratnayake A, Gomes G, Stoecker C, Kissinger PJ. Effectiveness of Incentivized Peer Referral to Increase Enrollment in a Community-Based Chlamydia Screening and Treatment Study Among Young Black Men. J Racial Ethn Health Disparities. 2024 Jun;11(3):1173-1181. doi: 10.1007/s40615-023-01595-5. Epub 2023 Apr 24. PMID 37095285